CLINICAL TRIAL: NCT02144480
Title: Efficacy of Early Short-term Training on Thrombogenesis in Patients Following Coronary Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 102-3049A3
Record Dates: First submitted 2014-05-01; First posted 2014-05-22 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-08

CONDITIONS: Coronary Artery Disease
Keywords: coronary bypass surgery; rehabilitation; exercise training; platelet activation; cardiopulmonary fitness
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive training (Experimental): intensive aerobic training in moderate intensity day5 postoperatively. 30 minutes per sessions, 2 sessions per day, 10 sessions per week. There will be 20 sessions in total.
  Interventions: Behavioral: Intensive training
- traditional training (Sham Comparator): traditional rehabilitation
  Interventions: Behavioral: traditional training

INTERVENTIONS:
Behavioral: Intensive training — The IT group will receive physiotherapy twice daily with longer duration and higher intensity
  Arms: Intensive training
Behavioral: traditional training — usual care: conventional rehabilitation
  Arms: traditional training

SUMMARY:
Although the benefit of cardiac rehabilitation following coronary artery bypass graft (CABG) is well-established, it is underused. The current investigation will adopt an early, intensive, short-term and supervised aerobic training at moderate-intensity. The inclusion criteria are diagnosed coronary artery disease (CAD) and clinical indication for elective first-time CABG.

Regular physical exercise is associated with overall reduced risk of primary cardiac arrest. Previous study demonstrated that moderate-intensity exercise training reduced resting and strenuous exercise-induced activation of platelet and possibly coagulation. Our main research question is that whether the short-term CR program in the present investigation will ameliorate hemostatic imbalance at rest and platelet coagulation activation at maximal stress exercise.

This is designed to be a prospective randomized controlled study. Sixty men who are scheduled to receive elective CABG in Chang Gung Memorial Hospital at Linkuo will be enrolled in the study. They will be randomized into two groups: intensive training (IT) and usual rehabilitation (UR). Participants in the IT group will receive intensive aerobic training at moderate intensity after CABG. A submaximal exercise test will be performed for intensity prescription. They will receive two training sessions per day and at least 20 sessions in total. The CR group will receive usual CR program. After intervention, each participant will receive a maximal exercise test. Additionally, six-minute walk test, generic and disease-specific quality of life, will be collected before and after training. Additional 20 age-matched non-sedentary and healthy men without training will be recruited as control group.

Venous blood will be sampled three times (before and after rehabilitation and maximal stress test) for the assessment of platelet activation by flow cytometer and activity of coagulation factors. Mean platelet volume, and platelet activation markers (platelet-bound CD62P%G, CD63%G, CD40L%G) will be analyzed. Various coagulation and fibrinolysis factors will be quantified.

We hypothesized that this training program will ameliorate the prothrombotic state and attenuate platelet reactivity and coagulation induced by strenuous exercise in patients after CABG. Hopefully, this clinical investigation will establish an early short-term rehabilitation model following CABG and its efficacy for clinical use.

DETAILED DESCRIPTION:
Introduction

The American College of Cardiology/American Heart Association guidelines suggested that cardiac rehabilitation (CR) should be offered to all eligible patients after coronary bypass surgery (CABG).[1] However, CR use in America is relatively low among Medicare beneficiaries despite convincing evidence of its benefits and recommendations for its use by professional organizations.[2] This neglect is as well evident in Taiwan. Traffic inconvenience and unavailability due to working hours are the common causes. There are ways to mend this situation. One of them is to develop an early, intensive and short-term CR program. The current investigation will adopt an early, intensive and supervised training for male patients following elective CABG due to old myocardial infarction and/or angina pectoris.

Meta-analyses of randomized controlled trials have consistently shown that participation in CR programs improves mortality and morbidity outcomes. It also benefits cardiopulmonary fitness, quality of life, lipid profile, etc.[3] Nonetheless, research regarding its effect on balance of thrombogenesis at rest or in response to vigorous exercise is either incomplete or controversial.

Previous studies found that acute physical exertion may trigger an acute coronary syndrome. The relative risk of cardiac events was 2-6 times higher during strenuous physical exertion (>6 METs) compared with during mild to moderate intensity activities in cardiac patients.[4] One of the possible explanations for this is that acute physical exertion may acutely change the hemostatic milieu in favor of increased coagulation and activation of platelet.[5] Available evidence suggests that strenuous exercise, in both healthy subjects and in various cardiovascular disease states, is associated with activation of platelets and blood coagulation, leading to a prothrombotic or hypercoagulable state.[6, 7] Aspirin is ineffective in attenuating enhanced platelet aggregation and activation induced by exercise.[8]

Regular physical exercise is associated with overall reduced risk of primary cardiac arrest.[4] D Wosornu et al. showed that a three-month aerobic training program (3 sessions per week) decreased resting fibrinogen concentration.[9] A meta-analysis showed that an exercise intervention over 2 weeks is associated with reduced inflammatory activity in patients with coronary artery disease (CAD). C-reactive protein and fibrinogen have provided the strongest evidence.[10] Platelet activation by strenuous exercise has been studied in 12 physically active and 12 sedentary individuals before and after a standardized treadmill exercise test. Among sedentary subjects, exercise caused an augmentation of the platelet activation and reactivity. In contrast, in physically active subjects exercise failed to induce alteration in platelet activation state.[11] Our previous study identified that moderate-intensity exercise training (60% maximal oxygen consumption for 30 min per day, 5 days/week for 8 weeks) reduced resting and strenuous exercise-induced platelet aggregation and platelet adhesion under shear flow in healthy men,[12] which were accompanied by decreased vWF binding to platelets and expression of P-selectin on platelets.[13] Accordingly, our main research question is that whether the short-term CR program in the current investigation ameliorates hemostatic imbalance at rest and platelet and coagulation activation at maximal stress exercise.

This is a prospective randomized controlled study. Sixty men who are scheduled to receive elective CABG in Chang Gung Memorial Hospital at Linkuo will be enrolled in the study. They will be randomized into two groups: intensive training (IT) and usual rehabilitation (UR). Participants in the IT group will receive education, reconditioning exercise and early intensive aerobic training at moderate intensity after CABG. A submaximal exercise test will be performed for prescription. They will receive two training sessions per day and at least 22 sessions in total. The CR group will receive usual CR program. After intervention, the participant will receive a maximal exercise test. In addition, six-minute walk test, generic and disease-specific quality of life will be collected before and after rehabilitation. Additional 20 age-matched, non-sedentary healthy participants without training will be recruited as control group.

Venous blood will be sampled three times (before and after rehabilitation and maximal stress test) for the assessment of platelet activation by flow cytometer and hemorheological profile by coagulation analyzer. Mean platelet volume, and platelet activation markers (platelet-bound CD62P%G, CD63%G, CD40L%G) will be analyzed. Various coagulation and fibrinolysis factors will be quantified including PT, aPTT, fibrinogen, thrombin time, FVIII:C, antithrombin, plasminogen, antiplasmin, anti-Xa and thrombin generation, D-Dimer, vWF etc.

We hypothesized that this training program will ameliorate the prothrombotic state and attenuate platelet reactivity and coagulation induced by strenuous exercise in patients after CABG. Hopefully, this clinical investigation will establish an early short-term rehabilitation model following CABG and its efficacy for clinical use.

Methodology

Participants A prospective study will be performed within the Cardiovascular Ward of Chang Gung Memorial Hospital, Linkuo. The inclusion criteria is diagnosed CAD and scheduled to receive elective CABG. Patients awaiting first-time elective CABG will be invited to participate in the study, and enrolled after giving written informed consent. Sixty patients will be enrolled. Exclusion criteria are musculoskeletal or neurological impairment precluding performance of cycling and walking assessment, atrial fibrillation, receiving anticoagulation therapy, inability to complete questionnaires, planned concomitant surgery, and a clinical status which requires emergent CABG. Additional 20 non-sedentary, age-matched healthy subjects without cardiovascular illness will be recruited as the control group. Non-sedentary life style is defined as walking more than 25 minutes in average per day according to the National Population Health Surveys of Canada. [14]

Randomization The patients will be randomized to two treatment groups (see Table 1 below) following assessment of study eligibility but prior to initial physiotherapy assessment. Randomization will be performed by means of random number generator based on their medical chart number. Thirty patients will be allocated to receive usual rehabilitation (UR); 30 to intensive training (IT).

Intervention protocol Physiotherapy interventions received by the two study groups are documented in Table 1. The IT group will receive physiotherapy twice daily with longer duration and higher intensity. After postoperative day5th, the training intensity will be prescribed at ventilatory anaerobic threshold (VAT) based on the submaximal exercise test in which the end point is supra-VAT. All physiotherapy interventions will be undertaken by one physiotherapist, specifically trained in the education and treatment methods used in the study.[15-17]

Supplemental oxygen will be used for all supervised/assisted walks if resting oxygen saturations is <92%. If patients are in sinus tachycardia (defined as >120 beats/min at rest) without hemodynamic compromise, exercise will be undertaken at a "comfortable" pace rather than at a "moderate" or "somewhat strong" level of perceived exertion. Patients will be counseled not to do walking training outside of physiotherapy sessions.

All patients will receive outcome assessment including cardiopulmonary exercise test, 6-minute-walk, quality of life, and hemorheological profile at basal and after strenuous exercise (Figure 1).

ELIGIBILITY:
Inclusion Criteria:

* CAD and scheduled to receive elective CABG. Male patients awaiting first-time elective CABG will be invited to participate in the study, and enrolled after giving written informed consent.

Exclusion Criteria:

* musculoskeletal or neurological impairment precluding performance of cycling and walking assessment
* receiving anticoagulation therapy
* inability to complete questionnaires
* a clinical status which requires emergent CABG
* end-stage renal disease
* peripheral arterial occlusive disease
* untreated life-threatening cardiac arrythmias
* acute heart failure
* uncontrolled hypertension
* advanced atrioventricular block
* acute myocarditis or pericarditis
* acute systemic illness
* intracardiac thrombus
* progressive worsening of exercise tolerance or dyspnea at rest over previous 3-5 days
* significant ischemia during low-intensity exercise (< 2 metabolic equivalent of tasks,< 50W)
* uncontrolled diabetes
* atrial fibrillation
* atrial flutter
* concurrent continuous or intermittent dobutamine therapy
* decrease in systolic blood pressure with exercise
* New York Heart Association (NYHA) class IV
* supine resting heart rate > 100 bpm

Ages: 20 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary fitness | 3 days to 4 weeks after coronary bypass
  before and after rehabilitation platelet activation before and after stress test

SECONDARY OUTCOMES:
platelet activity(composite measure) | 3 days to 4 weeks after coronary bypass
  by flow cytometry

OTHER OUTCOMES:
cardiovascular event | 3 weeks ~ 4 weeks s/p CABG
  acute myocardial infarction, hemodynamic instability during exercise training(SBP drop, ventricular tachycardia,...)

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Chun Huang, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Linkuo, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Woollard KJ, Geissmann F. Monocytes in atherosclerosis: subsets and functions. Nat Rev Cardiol. 2010 Feb;7(2):77-86. doi: 10.1038/nrcardio.2009.228. Epub 2010 Jan 12. PMID 20065951
- [Background] Geissmann F, Jung S, Littman DR. Blood monocytes consist of two principal subsets with distinct migratory properties. Immunity. 2003 Jul;19(1):71-82. doi: 10.1016/s1074-7613(03)00174-2. PMID 12871640
- [Background] Yang J, Zhang L, Yu C, Yang XF, Wang H. Monocyte and macrophage differentiation: circulation inflammatory monocyte as biomarker for inflammatory diseases. Biomark Res. 2014 Jan 7;2(1):1. doi: 10.1186/2050-7771-2-1. PMID 24398220
- [Background] Shantsila E, Wrigley B, Tapp L, Apostolakis S, Montoro-Garcia S, Drayson MT, Lip GY. Immunophenotypic characterization of human monocyte subsets: possible implications for cardiovascular disease pathophysiology. J Thromb Haemost. 2011 May;9(5):1056-66. doi: 10.1111/j.1538-7836.2011.04244.x. PMID 21342432
- [Background] Berg KE, Ljungcrantz I, Andersson L, Bryngelsson C, Hedblad B, Fredrikson GN, Nilsson J, Bjorkbacka H. Elevated CD14++CD16- monocytes predict cardiovascular events. Circ Cardiovasc Genet. 2012 Feb 1;5(1):122-31. doi: 10.1161/CIRCGENETICS.111.960385. Epub 2012 Jan 11. PMID 22238190
- [Background] Rogacev KS, Cremers B, Zawada AM, Seiler S, Binder N, Ege P, Grosse-Dunker G, Heisel I, Hornof F, Jeken J, Rebling NM, Ulrich C, Scheller B, Bohm M, Fliser D, Heine GH. CD14++CD16+ monocytes independently predict cardiovascular events: a cohort study of 951 patients referred for elective coronary angiography. J Am Coll Cardiol. 2012 Oct 16;60(16):1512-20. doi: 10.1016/j.jacc.2012.07.019. Epub 2012 Sep 19. PMID 22999728
- [Background] Ozaki Y, Imanishi T, Taruya A, Aoki H, Masuno T, Shiono Y, Komukai K, Tanimoto T, Kitabata H, Akasaka T. Circulating CD14+CD16+ monocyte subsets as biomarkers of the severity of coronary artery disease in patients with stable angina pectoris. Circ J. 2012;76(10):2412-8. doi: 10.1253/circj.cj-12-0412. Epub 2012 Jun 29. PMID 22785372
- [Background] Amir O, Spivak I, Lavi I, Rahat MA. Changes in the monocytic subsets CD14(dim)CD16(+) and CD14(++)CD16(-) in chronic systolic heart failure patients. Mediators Inflamm. 2012;2012:616384. doi: 10.1155/2012/616384. Epub 2012 Nov 27. PMID 23226928
- [Background] Vandendries ER, Furie BC, Furie B. Role of P-selectin and PSGL-1 in coagulation and thrombosis. Thromb Haemost. 2004 Sep;92(3):459-66. doi: 10.1160/TH04-05-0306. PMID 15351841
- [Background] Wrigley BJ, Shantsila E, Tapp LD, Lip GY. Increased formation of monocyte-platelet aggregates in ischemic heart failure. Circ Heart Fail. 2013 Jan;6(1):127-35. doi: 10.1161/CIRCHEARTFAILURE.112.968073. Epub 2012 Nov 14. PMID 23152489
- [Background] Michelson AD, Barnard MR, Krueger LA, Valeri CR, Furman MI. Circulating monocyte-platelet aggregates are a more sensitive marker of in vivo platelet activation than platelet surface P-selectin: studies in baboons, human coronary intervention, and human acute myocardial infarction. Circulation. 2001 Sep 25;104(13):1533-7. doi: 10.1161/hc3801.095588. PMID 11571248
- [Background] Czepluch FS, Kuschicke H, Dellas C, Riggert J, Hasenfuss G, Schafer K. Increased proatherogenic monocyte-platelet cross-talk in monocyte subpopulations of patients with stable coronary artery disease. J Intern Med. 2014 Feb;275(2):144-54. doi: 10.1111/joim.12145. Epub 2013 Oct 30. PMID 24118494
- [Background] Williams MA, Ades PA, Hamm LF, Keteyian SJ, LaFontaine TP, Roitman JL, Squires RW. Clinical evidence for a health benefit from cardiac rehabilitation: an update. Am Heart J. 2006 Nov;152(5):835-41. doi: 10.1016/j.ahj.2006.05.015. PMID 17070142
- [Background] Hubal MJ, Chen TC, Thompson PD, Clarkson PM. Inflammatory gene changes associated with the repeated-bout effect. Am J Physiol Regul Integr Comp Physiol. 2008 May;294(5):R1628-37. doi: 10.1152/ajpregu.00853.2007. Epub 2008 Mar 19. PMID 18353886
- [Background] Mikkelsen UR, Couppe C, Karlsen A, Grosset JF, Schjerling P, Mackey AL, Klausen HH, Magnusson SP, Kjaer M. Life-long endurance exercise in humans: circulating levels of inflammatory markers and leg muscle size. Mech Ageing Dev. 2013 Nov-Dec;134(11-12):531-40. doi: 10.1016/j.mad.2013.11.004. Epub 2013 Nov 25. PMID 24287006
- [Background] Lehmann M, Hasler K, Bergdolt E, Keul J. Alpha-2-adrenoreceptor density on intact platelets and adrenaline-induced platelet aggregation in endurance- and nonendurance-trained subjects. Int J Sports Med. 1986 Jun;7(3):172-6. doi: 10.1055/s-2008-1025757. PMID 3015811
- [Background] Adachi H, Itoh H, Sakurai S, Takahashi T, Toyama T, Naito S, Hoshizaki H, Oshima S, Taniguchi K, Kato M, Fu LT, Kato K. Short-term physical training improves ventilatory response to exercise after coronary arterial bypass surgery. Jpn Circ J. 2001 May;65(5):419-23. doi: 10.1253/jcj.65.419. PMID 11348046
- [Background] Mendes RG, Simoes RP, De Souza Melo Costa F, Pantoni CB, Di Thommazo L, Luzzi S, Catai AM, Arena R, Borghi-Silva A. Short-term supervised inpatient physiotherapy exercise protocol improves cardiac autonomic function after coronary artery bypass graft surgery--a randomised controlled trial. Disabil Rehabil. 2010;32(16):1320-7. doi: 10.3109/09638280903483893. PMID 20156053
- [Background] Hirschhorn AD, Richards D, Mungovan SF, Morris NR, Adams L. Supervised moderate intensity exercise improves distance walked at hospital discharge following coronary artery bypass graft surgery--a randomised controlled trial. Heart Lung Circ. 2008 Apr;17(2):129-38. doi: 10.1016/j.hlc.2007.09.004. Epub 2007 Dec 3. PMID 18060837
- [Background] Huang SC, Wong MK, Lin PJ, Tsai FC, Wen MS, Kuo CT, Hsu CC, Wang JS. Correction: Passive Leg Raising Correlates with Future Exercise Capacity after Coronary Revascularization. PLoS One. 2016 Jun 3;11(6):e0157205. doi: 10.1371/journal.pone.0157205. eCollection 2016. PMID 27257815
- [Background] Huang SC, Wong MK, Lin PJ, Tsai FC, Fu TC, Wen MS, Kuo CT, Wang JS. Modified high-intensity interval training increases peak cardiac power output in patients with heart failure. Eur J Appl Physiol. 2014 Sep;114(9):1853-62. doi: 10.1007/s00421-014-2913-y. Epub 2014 Jun 1. PMID 24880226
- [Background] Erratum: ATS Statement: Guidelines for the Six-Minute Walk Test. Am J Respir Crit Care Med. 2016 May 15;193(10):1185. doi: 10.1164/rccm.19310erratum. No abstract available. PMID 27174486
- [Background] Dill DB, Costill DL. Calculation of percentage changes in volumes of blood, plasma, and red cells in dehydration. J Appl Physiol. 1974 Aug;37(2):247-8. doi: 10.1152/jappl.1974.37.2.247. No abstract available. PMID 4850854
- [Background] Chen YC, Ho CW, Tsai HH, Wang JS. Interval and continuous exercise regimens suppress neutrophil-derived microparticle formation and neutrophil-promoted thrombin generation under hypoxic stress. Clin Sci (Lond). 2015 Apr;128(7):425-36. doi: 10.1042/CS20140498. PMID 25371035
- [Background] Fu TC, Wang CH, Lin PS, Hsu CC, Cherng WJ, Huang SC, Liu MH, Chiang CL, Wang JS. Aerobic interval training improves oxygen uptake efficiency by enhancing cerebral and muscular hemodynamics in patients with heart failure. Int J Cardiol. 2013 Jul 15;167(1):41-50. doi: 10.1016/j.ijcard.2011.11.086. Epub 2011 Dec 22. PMID 22197120
- [Background] Van Craenenbroeck AH, Van Ackeren K, Hoymans VY, Roeykens J, Verpooten GA, Vrints CJ, Couttenye MM, Van Craenenbroeck EM. Acute exercise-induced response of monocyte subtypes in chronic heart and renal failure. Mediators Inflamm. 2014;2014:216534. doi: 10.1155/2014/216534. Epub 2014 Dec 22. PMID 25587208
- [Background] Ahn KC, Jun AJ, Pawar P, Jadhav S, Napier S, McCarty OJ, Konstantopoulos K. Preferential binding of platelets to monocytes over neutrophils under flow. Biochem Biophys Res Commun. 2005 Apr 1;329(1):345-55. doi: 10.1016/j.bbrc.2005.01.146. PMID 15721313
- [Background] Burdess A, Nimmo AF, Campbell N, Harding SA, Garden OJ, Dawson AR, Newby DE. Perioperative platelet and monocyte activation in patients with critical limb ischemia. J Vasc Surg. 2010 Sep;52(3):697-703. doi: 10.1016/j.jvs.2010.04.024. PMID 20816321
- [Background] Lukasik M, Dworacki G, Kufel-Grabowska J, Watala C, Kozubski W. Upregulation of CD40 ligand and enhanced monocyte-platelet aggregate formation are associated with worse clinical outcome after ischaemic stroke. Thromb Haemost. 2012 Feb;107(2):346-55. doi: 10.1160/TH11-05-0345. Epub 2012 Jan 11. PMID 22234746
- [Background] Ardlie NG, Glew G, Schwartz CJ. Influence of catecholamines on nucleotide-induced platelet aggregation. Nature. 1966 Oct 22;212(5060):415-7. doi: 10.1038/212415a0. No abstract available. PMID 5970162
- [Background] Wang JS, Li YS, Chen JC, Chen YW. Effects of exercise training and deconditioning on platelet aggregation induced by alternating shear stress in men. Arterioscler Thromb Vasc Biol. 2005 Feb;25(2):454-60. doi: 10.1161/01.ATV.0000151987.04607.24. Epub 2004 Nov 29. PMID 15569820
- [Background] Shantsila E, Tapp LD, Wrigley BJ, Montoro-Garcia S, Ghattas A, Jaipersad A, Lip GY. The effects of exercise and diurnal variation on monocyte subsets and monocyte-platelet aggregates. Eur J Clin Invest. 2012 Aug;42(8):832-9. doi: 10.1111/j.1365-2362.2012.02656.x. Epub 2012 Feb 22. PMID 22356533
- [Background] Suaya JA, Shepard DS, Normand SL, Ades PA, Prottas J, Stason WB. Use of cardiac rehabilitation by Medicare beneficiaries after myocardial infarction or coronary bypass surgery. Circulation. 2007 Oct 9;116(15):1653-62. doi: 10.1161/CIRCULATIONAHA.107.701466. Epub 2007 Sep 24. PMID 17893274